CLINICAL TRIAL: NCT06420752
Title: Passive Stretching and Dietary Nitrate Rescue Functional Capacity in Peripheral Arterial Disease
Brief Title: Passive Stretching in Peripheral Arterial Disease Patients
Status: Recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: University of Wisconsin, La Crosse (Other)
Responsible Party: Principal Investigator, Jacob Caldwell, Assistant Professor, University of Wisconsin, La Crosse
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 232-JC-230.2
Record Dates: First submitted 2024-05-14; First posted 2024-05-20 (Actual); Last update posted 2025-04-02 (Actual); Status verified 2025-03

CONDITIONS: Peripheral Arterial Disease; Walking, Difficulty; Inflammation
Keywords: Cardiovascular
MeSH Terms: conditions — Peripheral Arterial Disease; Mobility Limitation; Inflammation

STUDY DESIGN:
Who Masked: Participant, Investigator
Masking Description: Double blind placebo controlled.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Functional Walking capacity (Experimental): Passive stretching of the calf muscles 5 days per week for 12-weeks
  Interventions: Device: Calf Plantar flexion; Dietary Supplement: Dietary nitrate
- Inflammation (Experimental): Blood and muscle biopsy samples pre/post passive stretching to assess local and systemic inflammation
  Interventions: Device: Calf Plantar flexion; Dietary Supplement: Dietary nitrate

INTERVENTIONS:
Device: Calf Plantar flexion — Daily passive calf stretching
Dietary Supplement: Dietary nitrate — Weekday 140 ml dietary nitrate consumption two hours prior to passive stretching

SUMMARY:
Peripheral artery disease (PAD) leads to higher mortality rates and strains healthcare systems due to increased costs. It causes leg pain during walking due to reduced blood flow. Nitric oxide (NO) deficiency contributes to vascular issues in PAD, with few effective treatments available. Passive calf muscle stretching boosts NO levels, vascular health, and walking ability in PAD patients. However, the inflammatory processes underlying these improvements are unclear. This study aims to track inflammatory markers and cardiovascular changes during 12 weeks of passive stretching. Additionally, combining stretching with dietary nitrate could further enhance walking capacity by reducing reactive oxygen species. The study will monitor inflammation, vascular function, and oxidative capacity to understand the effects on functional ability in PAD patients. This research is crucial for improving physical function and addressing exercise intolerance in PAD.

ELIGIBILITY:
Inclusion Criteria:

Ankle-brachial index of 0.90 or less Stable condition for at least 3 months

Exclusion Criteria:

Habitual exercise or cardiovascular rehabilitation program during the past 3 months Critical limb ischemia, amputation, or leg pain at rest Major surgery or lower extremity revascularization in the last 3 months Heart Failure Kidney disease Beet allergy Crohn's Current smoker

Ages: 40 Years to 90 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 64 (Estimated)
Dates: Start 2024-05-20 (Actual); Primary Completion 2028-12-31 (Estimated); Study Completion 2029-12-31 (Estimated)

PRIMARY OUTCOMES:
Functional capacity | 12-14 weeks
  6-minute walking distance will be assessed prior to an at various time points during the 12-week study

SECONDARY OUTCOMES:
Inflammatory markers | 12-14 weeks
  Blood and calf muscle biopsy will be used to assess various inflammatory markers pre/post treatment.
Vascular function | 12-14 weeks
  Large vessel (flow-mediated vasodilation) and small vessel (Near-infrared spectroscopy on the calf) will be measured prior to and at various time points during the 12-week study.

CONTACTS AND LOCATIONS:
Overall Officials: Jacob T Caldwell, Ph.D., Principal Investigator — Assistant Professor
Locations (1):
- University of Wisconsin La Crosse, La Crosse, Wisconsin, United States

IPD SHARING:
Plan to Share IPD: Yes
The study datasets will be submitted to a generalist repository (Aging Research Bio Bank or similar). This allows for individual-level data submission from clinical studies. This study will not generate genomics data and will not submit to the database of Genotypes and Phenotypes. To our understanding, the National Institutes of Aging repository is the only current general repository for aging related work
Supporting Information: Study Protocol, SAP, ICF
Time Frame: Raw data will be available after two years post data collection to allow for publication and only available for one year after data collection is complete.
Access Criteria: Researchers.

DOCUMENTS (2):
  • Study Protocol (2024-05-06): https://cdn.clinicaltrials.gov/large-docs/52/NCT06420752/Prot_000.pdf
  • Statistical Analysis Plan (2024-05-06): https://cdn.clinicaltrials.gov/large-docs/52/NCT06420752/SAP_001.pdf